CLINICAL TRIAL: NCT01241422
Title: A Randomized, Double-Blind, Placebo- and Active-Controlled Crossover Study to Evaluate the Efficacy of JNJ 40929837 for the Treatment of Asthma Using a Bronchial Allergen Challenge Model
Brief Title: A Study to Evaluate the Effectiveness of JNJ 40929837 for the Treatment of Asthma Using a Bronchial Allergen Challenge Model
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR017533; 40929837ASH2001 (Other: Johnson & Johnson Pharmaceutical Research and Development, L.L.C.)
Record Dates: First submitted 2010-10-25; First posted 2010-11-16 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-12

CONDITIONS: Asthma
Keywords: Asthma; Mild asthma; Singulair; JNJ 40929837; Montelukast
MeSH Terms: conditions — Asthma | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Treatment A: JNJ 40929837 (Experimental)
  Interventions: Drug: JNJ 40929837
- Treatment B: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Treatment C: Montelukast (Other)
  Interventions: Drug: Montelukast

INTERVENTIONS:
Drug: JNJ 40929837 — On Day 1: participants will receive 2 tablets of 50 mg JNJ 40929837 in the morning and 1 placebo capsule in the evening; from Days 2 to 6: they will receive 1 tablet of 50 mg JNJ 40929837 in the morning and 1 JNJ 40929837 50 mg tablet + 1 placebo capsule in the evening; and on Day 7: 1 tablet of 50 mg JNJ 40929837 in the morning.
  Arms: Treatment A: JNJ 40929837
Drug: Placebo — On Day 1: participants will receive 2 placebo tablets in the morning and 1 placebo capsule in the evening; from Days 2 to 6: they will receive 1 placebo tablet in the morning and 1 placebo tablet + 1 placebo capsule in the evening; and on Day 7: 1 placebo tablet in the morning.
  Arms: Treatment B: Placebo
Drug: Montelukast — On Day 1: participants will receive 2 placebo tablets in the morning and 1 montelukast capsule in the evening; from Days 2 to 6: they will receive 1 placebo tablet in the morning and 1 montelukast capsule + 1 placebo tablet in the evening; and on Day 7: 1 placebo tablet in the morning.
  Arms: Treatment C: Montelukast

SUMMARY:
The purpose of this study is to evaluate the allergen-induced late asthmatic response (LAR), as measured by maximal percent fall in forced expiratory volume in 1 second, in participants with stable mild atopic asthma after treatment with JNJ 40929837 as compared to placebo.

DETAILED DESCRIPTION:
This is a multicenter (study conducted at multiple sites), randomized (the study medication is assigned by chance), double-blind (neither the physician nor participant will know which of the treatments a participant is receiving, but can access the information in case of an emergency), and crossover (method used to switch participants from one treatment arm to another in a clinical study) study. Approximately 18 participants will participate in the study. The study will consist of screening phase (30 days before the administration of study drug), treatment phase, and follow-up phase (2 weeks after the end of the last treatment period). Participants will be randomly assigned to receive JNJ 40929837, placebo, and montelukast. Each participant will receive all the 3 treatments (7 days per treatment) and each treatment will be separated by 14 days of wash-out period (no treatment). Safety evaluations will include assessments of adverse events, clinical laboratory tests, electrocardiogram, vital signs, and physical examination, which will be evaluated throughout the study. The maximum study duration for a participant will be approximately 51 days.

ELIGIBILITY:
Inclusion Criteria: - Generally healthy - Have mild atopic asthma requiring no other treatment besides occasional short-acting beta-2-agonists - Have allergen-induced early asthmatic response of at least a 20 percent reduction in forced expiratory volume in 1 second (FEV1) and late asthmatic response of at least a 15 percent reduction in FEV1 during bronchial allergen challenge performed at screening - Females who are post menopausal, surgically sterilized, or practicing a highly effective method of birth control - Have an FEV1 at screening visit at least 75 percent of the predicted value - Have a history of asthma symptoms during exposure to indoor or outdoor allergens and a positive prick skin test done at the study site to dust mite, mixed grass pollen, or cat dander Exclusion Criteria: - Worsening of asthma or a respiratory tract infection within 6 weeks - HIV or Hepatitis B or C positive - Receipt of an investigational drug or use of an investigational medical device within the last month - Use of tobacco products of any kind currently or within 6 months - Have clinically significant abnormal physical examination, vital signs, or 12 lead electrocardiogram at screening as deemed appropriate by the investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2010-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Change in forced expiratory volume in 1 second (FEV1) during the late response to allergen | 3 to 10 hours after allergen exposure on Day 6 of each treatment period

SECONDARY OUTCOMES:
Change in FEV1 during the early response to allergen | 0-2 hours after allergen exposure on Day 6 of each treatment period
Area under the FEV1/time curve during the early response to allergen | Between 0 and 2 hours post allergen challenge on Day 6
Area under the FEV1/time curve during the late response to allergen | Between 3 and 10 hours post allergen challenge on Day 6
Plasma concentration of JNJ 40929837 | Day 1 (predose and 1, 2, 3, and 4 hours), pre-bronchial allergen challenge (BAC) Day 5 (predose and 2 hours), BAC Day 6 (predose and post-BAC [2 and 7 hours]), post-BAC Day 7 (predose and 2 hours), and follow-up visit
Sputum leukotriene B4 levels | Day 1 (predose and 2 and 4 hours), pre-BAC Day 5 (predose), BAC Day 6 (predose, post-BAC [2 and 7 hours]), post-BAC Day 7 (predose), and follow-up visit
  This biomarker will be measured as a pharmacodynamic evaluation.
Plasma leukotriene B4 levels | Day 1 (predose and 2 and 4 hours), pre-BAC Day 5 (predose), BAC Day 6 (predose, post-BAC [2 and 7 hours]), post-BAC Day 7 (predose), and follow-up visit
  This biomarker will be measured as a pharmacodynamic evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (2):
- Berlin, Germany
- Harrow, United Kingdom

REFERENCES:
- [Derived] Barchuk W, Lambert J, Fuhr R, Jiang JZ, Bertelsen K, Fourie A, Liu X, Silkoff PE, Barnathan ES, Thurmond R. Effects of JNJ-40929837, a leukotriene A4 hydrolase inhibitor, in a bronchial allergen challenge model of asthma. Pulm Pharmacol Ther. 2014 Oct;29(1):15-23. doi: 10.1016/j.pupt.2014.06.003. Epub 2014 Jul 10. PMID 25018015
- See also: Effects of JNJ-40929837, a leukotriene A4 hydrolase inhibitor, in a bronchial allergen challenge model of asthma W. 16 Barchuk et al. / Pulmonary Pharmacology & Therapeutics 29 (2014) 15e23 — http://dx.doi.org/10.1016/j.pupt.2014.06.003